CLINICAL TRIAL: NCT02031887
Title: Effect of a Starter Formula With Synbiotics on Stool Microbiota in Infants After Normal or Caesarean Section Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: South African Health Authorities now promote that HIV positive mothers should receive anti-retroviral drugs and breastfeed their infants.
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 07.19.INF
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Full Term Infants
Keywords: starter formula; stool microbiota; infants; caesarean section delivery
MeSH Terms: interventions — Food, Formulated; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infant starter formula with synbiotics (Experimental): Infant starter formula with synbiotics
  Interventions: Dietary Supplement: formula with synbiotics
- Infant formula without synbiotics (Active Comparator): Infant formula without synbiotics
  Interventions: Dietary Supplement: formula without synbiotics

INTERVENTIONS:
Dietary Supplement: formula with synbiotics
  Arms: Infant starter formula with synbiotics
Dietary Supplement: formula without synbiotics
  Arms: Infant formula without synbiotics

SUMMARY:
The primary objectives of this trial are:

* to show differences in the colonization of the gastrointestinal tract with the bacteria Bifidobacterium sp. between infants born by normal or caesarean delivery, fed with the test or a control product
* to investigate whether there is equivalence in growth between the four different groups of infant described above.

DETAILED DESCRIPTION:
The primary objectives of this trial are:

* to show differences in the colonization of the gastrointestinal tract with the bacteria Bifidobacterium sp. between infants born by normal or caesarean delivery, fed with the test or a control product
* to investigate whether there is equivalence in growth between the four different groups of infant described above.

Design:

This is a controlled, double blind, randomized, multi center, clinical trial of 4 groups in parallel.

Two groups of infants (born from normal or caesarean delivery) will each consume one of 2 milk formulae.

Number of patients (to be enrolled / to be analyzed): Approximately 450 / 240 Stratification will be done by gender and delivery mode.

Description of subjects and main criteria for inclusion:

Healthy full term infants born from HIV positive mothers who have elected to feed their child exclusively with a milk formula from birth. Children born after normal or caesarean delivery will be considered separately.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant from HIV positive mother
* Full term infant (more or equal to 37 weeks gestation; less or equal to 42 weeks gestation)
* Age of infant 3 days at the time of enrollment
* Birth weight between 2500 and 4500 grams
* Singleton birth
* The infant's mother has elected to feed their child exclusively with a milk formula from birth
* Informed consent from the parent or legal guardian

Exclusion Criteria:

* Congenital illness or malformation that may affect normal growth
* Significant pre-natal and / or post-natal disease
* Newborns who have received antibiotics during the first 3 days of life
* Newborns whose parents / caregivers cannot be expected to comply with the study protocol
* Newborns currently participating in another clinical trial

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2008-10; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
differences in the colonization of the gastrointestinal tract with the bacteria Bifidobacterium sp. between infants born by normal or caesarean delivery, fed with the test or a control product | 3 days, 10 days, 1 month, and 3 months of age of the infant
• Mean weight gain (g/day) | over 112 days

SECONDARY OUTCOMES:
body composition by DEXA | 4 month and 12 month of life
Digestive tolerance (stool characteristics and frequency, vomiting, regurgitation, frequency of colic) | 10 days, 1 month, 6 weeks, 3 month and 4 month of life

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Cooper, Principal Investigator — Witswatersrand University
Locations (3):
- South Africa (3):
  - Witswatersrand University, Johannesburg, Parktown
  - Chris Hani Baragwanath Hospital, Bertsham
  - Rahima Moosa Mother and Child Hospital, Johannesburg